CLINICAL TRIAL: NCT04132024
Title: Feasibility of Insomnia Tracking and Treatment in IBD (FITT)
Brief Title: Feasibility of Insomnia Tracking and Treatment in IBD
Acronym: FITT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Jessica.K.Salwen-Deremer, Assistant Professor, Departments of Psychiatry & Medicine, Section of Gastroenterology & Hepatology, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D19155
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Inflammatory Bowel Diseases; Insomnia
Keywords: Cognitive Behavioral Therapy for Insomnia (CBT-I); Insomnia; Sleep; Crohn's Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Sleep Initiation and Maintenance Disorders; Crohn Disease; Colitis, Ulcerative | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Behavioral Therapy for Insomnia (Experimental): CBT-I has a specific protocol with behavioral targets that differ significantly from standard CBT. This approach focuses on implementing sleep restriction and stimulus control interventions which are fully deployed during the first session. We will deliver 5 CBT-I sessions over the course of 8 weeks. Key recommendations include: 1) reduce time in bed; 2) get up at the same time every day; 3) do not go to bed unless sleepy; 4) do not stay in bed awake for more than 15 minutes; and 5) avoid napping. Participants are also taught relaxation strategies and cognitive therapy addresses arousal and catastrophizing.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I) — CBT-I has a specific protocol with behavioral targets that differ significantly from standard CBT. This approach focuses on implementing sleep restriction and stimulus control interventions which are fully deployed during the first session. 5 CBT-I sessions will be delivered over the course of 8 weeks. Key recommendations include: 1) reduce time in bed; 2) get up at the same time every day; 3) do not go to bed unless sleepy; 4) do not stay in bed awake for more than 15 minutes; and 5) avoid napping. Participants are also taught relaxation strategies and cognitive therapy addresses arousal and catastrophizing.

SUMMARY:
This study is a longitudinal clinical trial designed to characterize sleep patterns in individuals with Inflammatory Bowel Disease (IBD) as well as to assess the feasibility of sleep intervention (Cognitive Behavioral Therapy for Insomnia (CBT-I)) in individuals with both insomnia and Inflammatory Bowel Disease (IBD).

ELIGIBILITY:
Inclusion Criteria (IBD Participants):

* Documented IBD
* Mild to moderate Crohn's Disease or Ulcerative Colitis as measured by the Physicians Global Assessment

Inclusion Criteria (Healthy Participants)

* No personal history of IBD
* No personal history of Irritable Bowel Syndrome (IBS) or Celiac Disease
* No current gastrointestinal symptoms or concerns
* No family history of IBD or Celiac Disease

Exclusion Criteria (both IBD participants and healthy participants)

* PHQ-9 depression score > 15
* GAD-7 anxiety score > 15
* Current alcohol or substance abuse
* Current narcotic use
* Unstable major psychiatric condition
* Current sleep apnea or restless leg syndrome
* Other problems that would interfere with study participation at investigator discretion

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Change in sleep continuity | Tracking Study: Baseline (average of weeks 1 & 2), Treatment Study: Follow Up (change from baseline to week 15)
  Sleep continuity will be measured by sleep onset latency (SOL), wake after sleep onset (WASO), total sleep time (TST), and sleep efficiency (SE), based on ActiGraph data and daily diary data. Sleep parameters measured by the ActiGraph model wGT3X-BT, a wrist-accelerometer. Measured in minutes of sleep per night. Higher number indicating longer sleep duration.
Recruitment Rate | Tracking Study: Baseline (Week 1)
  Number of participants screened into the study per month will help measure feasibility.
Completion of Study Measures-Tracking Study | Baseline (average of weeks 1 & 2)
  The average percentage of study measures (daily diaries and CBT-I sessions) that are completed across participants will help determine feasibility.
Completion of Study Measures- Treatment Study | Follow Up (week 15)
  The average percentage of study measures (daily diaries and CBT-I sessions) that are completed across participants will help determine feasibility.
ActiGraph Use-Tracking Study | Baseline (Week 1)
  The average percentage of days spent wearing the medical-grade Fitbit-like-device that collects sleep and physical activity data to help assess feasibility.
ActiGraph Use-Treatment Study | Follow Up (week 15)
  The average percentage of days spent wearing the medical-grade Fitbit-like-device that collects sleep and physical activity data to help assess feasibility.
Actigraph Compliance-Tracking Study | Baseline (Week 1)
  The average percentage of hours of wear per day of the medical-grade Fitbit-like-device that collects sleep and physical activity data to help assess feasibility.
Actigraph Compliance-Treatment Study | Follow up (Week 15)
  The average percentage of hours of wear per day of the medical-grade Fitbit-like-device that collects sleep and physical activity data to help assess feasibility.

SECONDARY OUTCOMES:
Treatment liking | Treatment Study: Visit 1 (Week 3) and Follow up (Week 15)
  Treatment Acceptability Questionnaire will measure acceptability with patient-reported treatment satisfaction, and open-ended questions about satisfaction with both CBT-I and telemedicine (e.g., "What did you think about treating sleep as part of your IBD care?"; "How did you feel about getting treatment without being face-to-face?"; "What could we do to improve your treatment experience?").
Change in Sleepiness | Tracking Study: Baseline (Week 1) and Follow up (Week 15)
  The Epworth Sleepiness Scale will be used to assess general daytime sleepiness. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life, or their 'daytime sleepiness
Restless Leg Syndrome | Tracking Study: Baseline (Week 1)
  The Cambridge Hopkins Restless Leg Syndrome questionnaire will be used to assess the likelihood of Restless Leg Syndrome (RLS). Participants are categorized into definite not RLS, not RLS, probable RLS, and definite RLS based on item response patterns. A total score is not calculated.
Change in beliefs and attitudes about sleep | Tracking Study: Baseline (Week 1), Treatment Study: Visit 5 (Week 11), Follow up (Week 15)
  The Dysfunctional Beliefs & Attitudes About Sleep questionnaire will be used to assess beliefs about sleep. Except for item 23 (on the 30-item version) for which the score is reversed, a higher score indicates more dysfunctional beliefs and attitudes about sleep. The total score is based on the average score of all items. Subscale scores can be computed by adding the sum of scores for the items and dividing by the number of items making up each subscale.
Change in Insomnia Severity | Tracking Study: Baseline (Week1), Treatment Study: Visit 1 (Week 3), Visit 5 (Week 11) Follow up (Week 15)
  The Insomnia Severity Index will be used to assess insomnia symptoms. The total score ranges from 0 to 63, with higher scores indicating more severe anxiety symptoms.
Circadian Rhythms | Tracking Study: Baseline (Week 1)
  The Morningness-Eveningness Questionnaire (MEQ) will be used to assess whether the patient's circadian rhythm produces peak alertness in the morning or the evening. Multiple choice, 4-5 point scale. The sum gives a score ranging from 16 to 86; scores of 41 and below indicate "evening types", scores of 59 and above indicate "morning types", scores between 42-58 indicate "intermediate types".
Change in general fatigue | Tracking Study: Baseline (Week 1), Treatment Study: Follow up (Week 15)
  The Multidimensional Fatigue Inventory will be used to assess general fatigue. Items are scored 1-5, with 10 positively phrased items reverse scored (this concerns following items: 2, 5, 9, 10, 13, 14, 16, 17, 18, 19). For each of the 5 scales (general fatigue, physical fatigue, reduced activity, reduced motivation, and mental fatigue) a total score is calculated by summation of the scores of the individual items. Scores can range from the minimum of 4 to the maximum of 20.
Change in general sleep quality | Tracking Study: Baseline (Week 1), Treatment Study: Visit 1 (week 3), Visit 5 (week 11), Follow up (week 15)
  The Pittsburg Sleep Quality Index will be used to assess general sleep quality and disturbances. A total score of 5 or more is indicative of poor sleep quality. Possible score range is 0-21.
Change in behaviors that can interfere with sleep. | Tracking Study: Baseline (Week 1), Treatment Study: Visit 5 (Week 11), Follow up (week 15)
  The Sleep Hygiene Index will be used to assess the presence of behaviors that can interfere with sleep. A 13-item self-report measure designed to assess the practice of sleep hygiene behaviors. Each item is rated on a five-point scale ranging from 0 (never) to 4 (always). Total scores range from 0 to 52, with a higher score representing poorer sleep hygiene.
Sleep Apnea | Tracking Study: Baseline (Week 1)
  The STOP-BANG Questionnaire will be used to assess the patient's risk for sleep apnea. Scores range from 0-8. The higher the score indicates an increase in the probability of sleep apnea.
Change in pain | Tracking Study: Baseline (Week 1), Treatment Study: Visit 1 (week 3), Visit 5 (week 11), Follow up(week 15)
  The Brief Pain Inventory will be used to assess pain location, severity, and interference. Pain severity is rated from 0-10 and pain interference is rated from 0-10; higher scores indicate more severe pain and more pain interference.
Change in pain related disability | Tracking Study: Baseline (Week 1), Follow up (Week 15)
  The Graded Chronic Pain Scale will be used to assess the pain-related disability. Responses are translated into a chronic pain grade, from 0 (no pain) to 4 (severe interference).
Change in beliefs about pain | Tracking: Baseline (Week 1), Follow up (week 15)
  The Pain Catastrophizing Scale will be used to assess beliefs about pain. Scores range from 0-52, with higher scores indicating greater catastrophizing.
Change in individual's beliefs about IBD symptoms | Tracking Study: Baseline (Week 1), Treatment: Visit 1 (week 3), Visit 5 (week 11), Follow up (week 15)
  The Overall Disease Severity Index will be used to assess an individual's beliefs about IBD symptoms. This is a single item measure, with higher scores indicating greater IBD severity.
Change in IBD severity | Tracking Study: Baseline (Week 1), Treatment: Visit 1 (week 3), Visit 5 (week 11), Follow up (week 15)
  The Physicians Global Assessment will be used to complete a physician rated IBD severity assessment; physicians categorize severity of IBD based on symptom presentation.
Change in IBD symptom severity | Tracking Study: Baseline (Week 1), Treatment: Visit 1 (week 3), Visit 5 (week 11), Follow up (week 15)
  Patient Reported Outcome Measures (PRO-3) will be used to assess the severity of IBD symptoms, where greater scores indicate more severe IBD symptoms.
Change in severity of anxiety symptoms | Tracking Study: Baseline (Week 1), Treatment Study: Visit 1 (week 3), Follow up (week 15)
  The Generalized Anxiety Disorder-7 will be used to assess overall severity of anxiety symptoms The GAD7 scores range from 5-21, with 5-9 indicating mild, 10-14 moderate, and greater than 15 severe anxiety.
Change in severity of depression symptoms | Tracking Study: Baseline (Week 1), Treatment Study: Visit 1 (week 3), Follow up (week 15)
  The Patient Health Questionnaire-9 will be used to assess overall severity of depression symptoms. The PHQ9 scores range from 0-27, with lower numbers indicating minimal to no depression and higher numbers indicating severe depression.
Change in stress | Tracking Study: Baseline (Week 1), Treatment Study: Follow up (week 15)
  The Perceived Stress Scale will be used to assess general stress. Individual scores can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress
Change in overall health and quality of life | Tracking Study: Baseline (Week 1), Treatment Study: Follow up (week 15)
  The Short Form-36 will be used to assess overall health and impact on quality of life. Consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] Salwen-Deremer JK, Reid MJ, Westvold SJ, Siegel CA, Smith MT. People with IBD evidence more microarousals during sleep architecture assessments. BMJ Open Gastroenterol. 2023 Dec 28;10(1):e001249. doi: 10.1136/bmjgast-2023-001249. PMID 38154825
- [Derived] Salwen-Deremer JK, Smith MT, Aschbrenner KA, Haskell HG, Speed BC, Siegel CA. A pilot feasibility trial of cognitive-behavioural therapy for insomnia in people with inflammatory bowel disease. BMJ Open Gastroenterol. 2021 Dec;8(1):e000805. doi: 10.1136/bmjgast-2021-000805. PMID 34969664